CLINICAL TRIAL: NCT05380635
Title: Phase 2a Study of Systemic PK and Serial ECG Determinations Following 8 Weeks of HyBryte Treatment
Brief Title: PK and ECG Determinations Following 8 Weeks of HyBryte Treatment for Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HPN-CTCL-02
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
Keywords: CTCL; MF; Hypericin; HyBryte
MeSH Terms: conditions — Mycosis Fungoides | interventions — hypericin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HyBryte (0.25 % Hypericin) (Experimental): HyBryte (0.25 % hypericin) ointment will be applied to CTCL lesions and treated with visible light 18-24 hours later starting at 5 J/cm^2. Drug application/light session will be done twice a week (at least 2 calendar days apart) for 8 weeks.
  Interventions: Drug: Hypericin

INTERVENTIONS:
Drug: Hypericin — HyBryte is synthetic hypericin formulated as a 0.25% hypericin ointment.
  Other Names: HyBryte; SGX301

SUMMARY:
To assess the blood levels of hypericin and any electrocardiogram (ECG) changes during 8 weeks of HyBryte (topical hypericin ointment) photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of cutaneous T-cell lymphoma (CTCL, mycosis fungoides), Stage IB or Stage IIA
* CTCL lesions covering ≥ 10% of their body surface area

Exclusion Criteria:

* History of allergy or hypersensitivity to any of the components of HyBryte
* Pregnancy or mothers who are breast-feeding
* Males and females not willing to use effective contraception
* Subjects with history of sun hypersensitivity or photosensitive dermatoses (e.g., porphyria, systemic lupus erythematosus (SLE), Sjogren's syndrome, etc.)
* Subjects whose condition is spontaneously improving
* Subjects receiving topical steroids or other topical treatments (e.g., nitrogen mustard) on index lesions for CTCL within 2 weeks of enrollment
* Subjects receiving systemic steroids, psoralen ultraviolet A (UVA) radiation therapy (PUVA), narrow band ultraviolet B (UVB) light therapy (NB-UVB) or carmustine (BCNU) or other systemic therapies for CTCL within 3 weeks of enrollment
* Subjects who have received electron beam irradiation within 3 months of enrollment
* Subjects with a history of significant systemic immunosuppression
* Subjects taking other investigational drugs or drugs of abuse within 30 days of enrollment
* Subjects receiving drugs known to cause photosensitization within 2 weeks of starting HyBryte therapy unless they have not had evidence of photosensitization after receiving a stable dose of the medication for a minimum of 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Skin Lymphoma Medical Group, Fairport, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HyBryte (0.25 % Hypericin)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Electrocardiograms (ECG)
Description: Assess any ECG QT interval changes (defined as any occurrences of QT interval >500 ms or changes in QT interval >60 ms) during standard HyBryte photodynamic therapy.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Systemic Blood Levels
Description: Assess the systemic blood levels of hypericin during standard HyBryte photodynamic therapy.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
ug/mL | 0.00013 (0.00011)

3. Secondary Outcome: Number of Responders and Non-Responders With a Treatment Response in 3 Treated Lesions as Defined as a ≥50% Improvement in the Composite Assessment of Index Lesion Disease Severity (CAILS) Score.
Description: A treatment response was defined as a ≥50% improvement in CAILS score at Week 10 when compared to the CAILS score at baseline.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
  The overall CAILS score was calculated by adding the total score as described above for each of the 3 lesions. The overall CAILS score has a range of 0 to 111. A lower score means a better outcome.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
Participants
  Responder | 2
  Non-Responder | 7

4. Secondary Outcome: Number of Index Lesions With a Treatment Response as Defined as a ≥50% Improvement in the Composite Assessment of Index Lesion Disease Severity (CAILS) Score.
Description: A treatment response was defined as a ≥50% improvement in CAILS score at Week 10 when compared to the CAILS score at baseline in each of the individual Index Lesions.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
Time Frame: 10 weeks
Population: Each participant had 3 Index Lesions treated and evaluated
Measure: Count of Units; unit: Index Lesions
Units Other Than Participants: Index Lesions
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
Number analyzed (Index Lesions) | 27
Index Lesions
  Responder | 7
  Non-Responder | 20

5. Secondary Outcome: Number of Index Lesions With a Complete Response as Defined as a 100% Improvement in the Composite Assessment of Index Lesion Disease Severity (CAILS) Score.
Description: A complete response was defined as a 100% improvement in CAILS score (a CAILS score of 0) at Week 10 in each of the individual Index Lesions.
  The Composite Assessment of Index Lesion Disease Severity (CAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
Time Frame: 10 weeks
Population: Each participant had 3 Index Lesions treated and evaluated
Measure: Count of Units; unit: Index Lesions
Units Other Than Participants: Index Lesions
Arm/Group | HyBryte (0.25 % Hypericin)
Number analyzed (Participants) | 9
Number analyzed (Index Lesions) | 27
Index Lesions
  Responder | 4
  Non-Responder | 23

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | HyBryte (0.25 % Hypericin)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HyBryte (0.25 % Hypericin) (N=9)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Chills (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT05380635/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT05380635/SAP_001.pdf